CLINICAL TRIAL: NCT04991155
Title: Effect of Food on BIA 5-1058 Bioavailability in Healthy Subjects
Brief Title: Effect of Food on BIA 5-1058
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-102; 2015-001951-65 (EudraCT Number)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PART 1 (400 mg BIA 5-1058) (Experimental): Each subject was orally administered a single oral dose of BIA 5-1058 on D1 (dosing day) on three different occasions (Period 1, Period 2 and Period 3): Part 1: 400 mg BIA 5-1058 as four (4) 100 mg tablets in Period 1, 400 mg BIA 5-1058 as four (4) 100 mg tablets in Period 2, and 400 mg BIA 5-1058 as four (4) 100 mg tablets in Period 3.
  Interventions: Drug: BIA 5-1058
- PART 2 (800 mg BIA 5-1058) (Experimental): Each subject was orally administered a single oral dose of BIA 5-1058 on D1 (dosing day) on three different occasions (Period 1, Period 2 and Period 3):
  Part 2: 800 mg BIA 5-1058 as eight (8) 100 mg tablets in Period 1, 800 mg BIA 5-1058 as eight (8) 100 mg tablets in Period 2, and 800 mg BIA 5-1058 as eight (8) 100 mg tablets in Period 3.
  Interventions: Drug: BIA 5-1058
- PART 3 (1200 mg BIA 5-1058) (Experimental): Each subject was orally administered a single oral dose of BIA 5-1058 on D1 (dosing day) on three different occasions (Period 1, Period 2 and Period 3):
  Part 3: 1200 mg BIA 5-1058 as twelve (12) 100 mg tablets in Period 1, 1200 mg BIA 5-1058 as twelve (12) 100 mg tablets in Period 2, and 1200 mg BIA 5-1058 as twelve (12) 100 mg tablets in Period 3.
  Interventions: Drug: BIA 5-1058

INTERVENTIONS:
Drug: BIA 5-1058 — BIA 5-1058 (tablets 100 mg) was administered orally with 240 mL (Part 1) or 270 mL (Part 2 and Part 3) of water, in one period in the morning under fasting conditions (after at least a 10-hour overnight fast), in one period in the morning after a moderate meal, and in the other period at lunch after a moderate meal.
  Other Names: Zamicastat

SUMMARY:
The aim of this study is to investigate the effect of food on the pharmacokinetic (PK) profile of BIA 5-1058 after a single dose in healthy subjects.

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, single-dose, three-way crossover, three-part study in 54 healthy subjects.

Duration of treatment:

The study comprised a screening evaluation between 2 and 28 days before the first IMP (Investigational Medicinal Product) administration and 3 treatment periods of approximately 4 days, separated by wash-out periods of at least 7 days. A follow-up visit was performed approximately 7 days after discharge from the last period or early discontinuation. For each subject, the full duration of the participation in the study was approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent and to comply with the study restrictions;
2. Male or female subjects aged 18 to 45 years, inclusive;
3. Body mass index (BMI) between 18 and 30 kg/m2, inclusive;
4. Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead electrocardiogram (ECG);
5. Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibodies (HCV Ab) and anti-human immunodeficiency virus antibodies (HIV-1 and HIV-2 Ab) at screening;
6. Clinical laboratory test results clinically acceptable at screening and admission to each treatment period;
7. Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period;
8. Non-smokers or ex-smokers for at least 3 months.

   If female:
9. No childbearing potential by reason of surgery or at least 1 year post menopause (i.e., 12 months post last menstrual period), or menopause confirmed by follicle-stimulating hormone (FSH) testing;
10. If of childbearing potential, she was using an effective non-hormonal method of contraception [intrauterine device or intrauterine system; condom or occlusive cap (diaphragm or cervical or vault caps) with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he is the sole partner of that subject] for all the duration of the study;
11. Negative serum pregnancy test at screening and negative urine pregnancy test on admission of each treatment period (women of childbearing potential only).

    If male:
12. Using an effective method of contraception with a pregnant partner or partner of childbearing potential (condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomy) throughout the study;
13. Refraining from donating sperm throughout the study.

Exclusion Criteria:

1. Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders;
2. Clinically relevant surgical history;
3. History of relevant atopy or drug hypersensitivity;
4. History of alcoholism or drug abuse;
5. Consumption of more than 14 units of alcohol a week [1 glass (25 cL) of beer with 3° of alcohol = 7.5 g, or 1 glass (25 cL) of beer with 6° of alcohol = 15 g, or 1 glass (12.5 cL) of wine with 10° of alcohol = 12 g, or 1 glass (4cL) of aperitif with 42° of alcohol = 17 g];
6. Significant infection or known inflammatory process at screening or admission to each treatment period;
7. Display of acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period;
8. Use of medicines within 2 weeks of admission to the first period that may could affect the safety or other study assessments, in the Investigator's opinion;
9. Previous administration of BIA 5-1058;
10. Use of any investigational drug or participation in any clinical trial within 90 days prior to screening;
11. Participation in more than 2 clinical trials within the 12 months prior to screening;
12. Donation or reception of any blood or blood products within the 3 months prior to screening;
13. Vegetarians, vegans or had any other medical dietary restrictions;
14. Not able to communicate reliably with the Investigator;
15. Unlikely to co-operate with the requirements of the study.

    If female:
16. Pregnant or breastfeeding;
17. Not using an accepted effective contraceptive method or was using oral contraceptives.

    If male:
18. Not using an accepted effective method of contraception;
19. Refusing to refrain from donating sperm throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 9 weeks
  In all treatment periods, blood samples were taken at the following times: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose
Time of occurrence of Cmax (tmax) | Up to 9 weeks
  In all treatment periods, blood samples were taken at the following times: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose
Area under the plasma concentration-time curve (AUC) | Up to 9 weeks
  In all treatment periods, blood samples were taken at the following times: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose
Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which the drug concentration was at or above the lower limit of quantification (AUC0-last) | Up to 9 weeks
  In all treatment periods, blood samples were taken at the following times: before BIA 5-1058 dosing, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose

IPD SHARING:
Plan to Share IPD: No